CLINICAL TRIAL: NCT01369173
Title: Metabolic Response to Western vs. Indigenous Diets in Hispanic Women
Brief Title: COMIDAS Comparing Original Mexican Diets and Standard US Diets
Acronym: COMIDAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: FHCRC IR 7099; P50CA148143 (NIH)
Record Dates: First submitted 2011-06-03; First posted 2011-06-08 (Estimated); Last update posted 2015-05-06 (Estimated); Status verified 2015-05

CONDITIONS: Healthy
Keywords: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mexican Menu (Active Comparator): 24 days, all foods and drinks provided, menu consists of traditional mexican meals
  Interventions: Other: Mexican or American foods
- US diet (Active Comparator): 24 days, all foods and drinks provided, menu consists of foods commonly eaten in contemporary United States
  Interventions: Other: Mexican or American foods

INTERVENTIONS:
Other: Mexican or American foods — Participants will be randomized to an isocaloric Indigenous Mexican or a Western diet for 24 days. All foods and beverages will be prepared by the Human Nutrition Laboratory at the Fred Hutchinson Cancer Research Center. After a 4-week wash-out period, participants will cross over to the other arm and be given the alternate diet for 24 days. Blood and urine specimens will be collected before and after each feeding period to test baseline and post-intervention metabolic response as defined by various inflammatory and cancer susceptibility biomarkers including insulin-like growth factor 1 (IGF1), insulin-like growth factor binding protein 3 (IGFBP3), leptin, adiponectin, interleukin-6 (IL-6), C-reactive protein (CRP) and SAA (serum amyloid-A). DNA extracted from whole blood will be used to test whether a panel of 128 Ancestry Informative Markers (AIMs) is associated with metabolic response to the diets and other phenotypic traits of obesity, which relate to breast cancer risk.

SUMMARY:
The foods eaten daily are considered the "dietary pattern" of a culture or country. The dietary pattern of Mexico is different from that of the United States. To look at the effects of these patterns, participants in this study eat a Mexican menu for three and a half weeks and an American menu for the same length of time. At the beginning and end of each menu period participants provide blood and urine samples which we analyze to compare the effects of each diet. More info at www.ProyectoCOMIDAS.info

DETAILED DESCRIPTION:
Chronic disease risk, including breast cancer risk, is not uniform across race and ethnic groups in the United States. This variation in disease risk may be due to environmental exposures (including diet), genetic susceptibility, disparities in access to health screening, diagnosis and medical care, or combination of these factors. Here we have shown that Hispanic women in the U.S. are more likely to be overweight or obese compared to non-Hispanic whites. Some of the excess obesity risk is likely due to the lack of neighborhood availability and affordability of fruit, vegetables, lean protein and whole grains. Whether an inexpensive and widely available highly processed/refined, nutrient poor diet superimposed on a genetic background favoring adipose deposition (i.e., the "thrifty genotype") is metabolically detrimental has not been investigated. Research to test the metabolic response to Indigenous and Western diets in Hispanic women may provide important information about the etiology of obesity and obesity-related diseases in Hispanic women, including risk of breast cancer. Since reducing disparities in obesity-related diseases, including breast cancer, is an important public health goal, identifying potential programs for prevention should receive high priority.

Mexicans are the largest immigrant group in the United States with an estimated 10 million Mexican-American women currently in the U.S. As they acculturate to this country, Mexican immigrants change their dietary habits from traditional (indigenous) foods with plentiful fruit, vegetables and complex carbohydrates rich in fiber and other compounds to a Western-style diet high in fat and refined carbohydrate, but low in plant foods. Particularly concerning is that the food choices made by Mexican immigrants, many of whom are of lower socio-economic status, are driven partly by their inability to procure and purchase healthy foods. The disparity in both food availability and purchasing power fuels a tendency to obtain and consume a low-cost, Western style diet. When this diet is superimposed on persons with a "thrifty genotype" who are evolutionarily adapted to diets high in legumes and complex carbohydrates, it may lead to an abnormal metabolic response that favors adipose deposition and numerous health risks. Thus, ancestral genetic characteristics likely have an important role in metabolic response to specific dietary patterns and subsequent health risks. This phenomenon may partly explain the tendency for Mexicans and other immigrants from the Americas to become obese after just one generation in the United States.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Women of Mexican Descent
* Age between 18-45 years

Exclusion Criteria:

1. current physician-diagnosed diseases that require dietary restrictions or certain medications, including but not limited to, diabetes mellitus, kidney disease, other metabolic disorders, and cardiovascular disease requiring diet modifications
2. impaired glucose tolerance defined as fasting glucose > 100 mg/dL; all participants will complete a fasting blood glucose determination
3. BMI < 18.5 kg/m2 or > 40.0 kg/m2
4. current pregnancy or pregnancy in last year, lactation or plans to become pregnant during the study period
5. cessation of menses (either natural or surgical)
6. any previous cancer diagnosis or treatment within the previous five years (excluding non-melanomatous skin cancer)
7. restrained eating habits
8. current use of tobacco (any smoking) or alcohol (> 2 drinks/day)
9. inability (e.g., food allergy/intolerances) or unwillingness to consume the study foods.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2011-10; Primary Completion 2014-08 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
metabolic response measured by blood concentrations of biomarkers | Change from Baseline at 24 days
  Participants will have a blood draw at the beginning and end of each intervention arm.

CONTACTS AND LOCATIONS:
Locations (1):
- Fred Hutchinson Cancer Research Center, Seattle, Washington, United States

REFERENCES:
- [Derived] Santiago-Torres M, De Dieu Tapsoba J, Kratz M, Lampe JW, Breymeyer KL, Levy L, Song X, Villasenor A, Wang CY, Fejerman L, Neuhouser ML, Carlson CS. Genetic ancestry in relation to the metabolic response to a US versus traditional Mexican diet: a randomized crossover feeding trial among women of Mexican descent. Eur J Clin Nutr. 2017 Mar;71(3):395-401. doi: 10.1038/ejcn.2016.211. Epub 2016 Dec 14. PMID 27966572
- [Derived] Santiago-Torres M, Kratz M, Lampe JW, Tapsoba Jde D, Breymeyer KL, Levy L, Villasenor A, Wang CY, Song X, Neuhouser ML. Metabolic responses to a traditional Mexican diet compared with a commonly consumed US diet in women of Mexican descent: a randomized crossover feeding trial. Am J Clin Nutr. 2016 Feb;103(2):366-74. doi: 10.3945/ajcn.115.119016. Epub 2015 Dec 30. PMID 26718418